CLINICAL TRIAL: NCT04508322
Title: Early and Late Treatment of Class II Malocclusion With Excessive Overjet- a Randomized Controlled Trial Regarding Treatment Results, Patient Experience and Treatment and Cost-effectiveness
Brief Title: Treatment of Class II Malocclusion With Excessive Overjet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jenny Kallunki (Other)
Collaborators: Region Östergötland (Other); Malmö University (Other); Eklund foundation Malmö (Unknown); Swedish Dental Associations Scientific Funds (Unknown)
Responsible Party: Sponsor-Investigator, Jenny Kallunki, Senior Consultant Orthodontist. PhD-student, Region Östergötland
Organization: Region Östergötland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Treatment of Class II maloccl.
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-04

CONDITIONS: Class II Malocclusion, Division 1; Orthodontic Appliances; Quality of Life; Costs and Cost Analysis
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Early treatment HGA (9 years)
  Interventions: Device: HGA; Device: FA
- Group 2 (Active Comparator): Late treatment HGA (11 years)
  Interventions: Device: HGA; Device: FA
- Group 3 (Active Comparator): Treatment FA
  Interventions: Device: FA

INTERVENTIONS:
Device: HGA — Headgear Activator
  Arms: Group 1; Group 2
Device: FA — Fixed Orthodontic Appliance

SUMMARY:
Class II malocclusion with excessive overjet is one of the most common malocclusions among children and adolescents. The overall goal of the project is to analyze orthodontic treatment of Class II malocclusion with excessive overjet when the treatment is started in different ages and treated with removable and/or fixed appliance.

Treatment initiated before the age of eleven is performed with a removable functional appliance, Headgear Activator (HGA). Treatment starting in early adolescence is performed with fixed orthodontic appliance (FA).

The hypotheses are:

* Treatment with HGA at the age of nine or eleven is effective. No spontaneous correction of the malocclusion is expected in the untreated control group.
* Patient experience, treatment effect and cost-effectiveness are equivalent whether the treatment with HGA is initiated at the age of nine or eleven.
* Treatment results, patient experience and treatment- and cost-effectiveness are equivalent whether treatment is initiated early with HGA or initiated in early adolescence with FA.
* The treatment of Class II malocclusion with excessive overjet renders long-term treatment stability and patient satisfaction.

DETAILED DESCRIPTION:
Participants (children, 9 years of age) are recruited at the orthodontic specialist clinic in Norrköping, Sweden.

After informed consent participants are randomized into Group 1, 2 or 3. After randomization and registration, treatment with HGA is initiated for Group 1.

Group 2 and 3 serves as untreated control group. Two years after registration, Group 2 starts treatment with HGA at the age of eleven.

Group 3 serves as untreated control group to treatment with HGA.

Four years after registration, Group 3 starts treatment with FA (3M Victory brackets, .022 slot size, McLaughlin-Bennet-Trevesi prescription).

The patients in group 1 and 2 in need of a second phase of orthodontic treatment are treated with FA (3M Victory brackets, .022 slot size, McLaughlin-Bennet-Trevesi prescription) in early adolescence.

The following registrations are made:

Study models, photographs (extraoral, intraoral), Lateral head radiographs (T0, T2, T5, if required T1, T3), Child perceptions questionnaire.

T0: After randomization; before treatment start (Group 1), registration/control (Group 2,3).

T1: Two years after T0; after finished treatment for (Group 1), before treatment start (Group 2), control/registration for (Group 3).

T2: Two years after T1; follow up (Group 1), after finished treatment (Group 2), before treatment start (Group 3).

T3: Approx two years after T2 for patients not undergoing treatment with FA. For patients treated with FA, when treatment is finished.

T4: Approx two years after T3- follow up.

T5: Approx 8-10 years after T0 (Long term follow-up)

ELIGIBILITY:
Inclusion Criteria:

* Eight to ten years of age at the start of the trial
* mixed dentition;
* Excessive overjet (≥ 6 mm) and first maxillary permanent molars in Class II malocclusion
* No sucking habits or ceased sucking habits should have been evident at least one year before the trial was started.

Exclusion Criteria:

* Craniofacial syndromes
* Previous orthodontic treatment
* Severe crowding of teeth, i.e. making the extraction of teeth necessary

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in overjet; i.e change in tooth position during treatment. Assessment at follow up. | Through study completion (T0-T5), an average of two years between controls.
  Tooth movement is assessed in millimeters by measures on study models.

SECONDARY OUTCOMES:
Change in Oral health related quality of life (OHRQoL) | Through study completion (T0-T5), an average of two years between controls.
  Oral health related quality of life is assessed by the use of the Child Perceptions Questionnaire where 0 is minimal and 148 is maximum. Higher scores corresponds to poorer OHRQoL.
Societal costs | During active treatment (T0-T3).
  Societal costs are the sum of indirect and direct treatment costs. Indirect treatment costs are travel costs for the patient and cost for parents when accompaning patients during treatment. Direct costs are clinical costs due to personnel and material.
Change in tooth position and skeletal growth. | Through study completion (T0-T5), an average of two years between controls.
  Tooth movement is assessed in millimeters by measures on study models. Skeletal growth is assessed in length and angular measures by cephalometric analysis of lateral radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Kallunki, Orthodontist, Principal Investigator — Malmö University
Locations (1):
- The Center for Orthodontics and Pedodontics, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spandrio L. [Pre-analysis variability: the effect of evaporation on the error of measurement, with special reference to sodium and potassium]. Quad Sclavo Diagn. 1984 Mar;20(1):110-21. Italian. PMID 6494411
- [Background] Dimberg L, Arnrup K, Bondemark L. The impact of malocclusion on the quality of life among children and adolescents: a systematic review of quantitative studies. Eur J Orthod. 2015 Jun;37(3):238-47. doi: 10.1093/ejo/cju046. Epub 2014 Sep 11. PMID 25214504
- [Background] Kallunki J, Sollenius O, Paulsson L, Petren S, Dimberg L, Bondemark L. Oral health-related quality of life among children with excessive overjet or unilateral posterior crossbite with functional shift compared to children with no or mild orthodontic treatment need. Eur J Orthod. 2019 Mar 29;41(2):111-116. doi: 10.1093/ejo/cjy033. PMID 29878165
- [Background] O'Brien K, Wright J, Conboy F, Chadwick S, Connolly I, Cook P, Birnie D, Hammond M, Harradine N, Lewis D, McDade C, Mitchell L, Murray A, O'Neill J, Read M, Robinson S, Roberts-Harry D, Sandler J, Shaw I, Berk NW. Effectiveness of early orthodontic treatment with the Twin-block appliance: a multicenter, randomized, controlled trial. Part 2: Psychosocial effects. Am J Orthod Dentofacial Orthop. 2003 Nov;124(5):488-94; discussion 494-5. doi: 10.1016/S0889540603006425. PMID 14614414
- [Background] Jokovic A, Locker D, Tompson B, Guyatt G. Questionnaire for measuring oral health-related quality of life in eight- to ten-year-old children. Pediatr Dent. 2004 Nov-Dec;26(6):512-8. PMID 15646914
- [Background] Jokovic A, Locker D, Stephens M, Kenny D, Tompson B, Guyatt G. Validity and reliability of a questionnaire for measuring child oral-health-related quality of life. J Dent Res. 2002 Jul;81(7):459-63. doi: 10.1177/154405910208100705. PMID 12161456
- [Background] Kallunki J, Bondemark L, Paulsson L. Early headgear activator treatment of Class II malocclusion with excessive overjet: a randomized controlled trial. Eur J Orthod. 2021 Dec 1;43(6):639-647. doi: 10.1093/ejo/cjaa073. PMID 33274388
- [Background] Kallunki J, Bondemark L, Paulsson L. Comparisons of costs and treatment effects-an RCT on headgear activator treatment of excessive overjet in the mixed and late mixed dentition. Eur J Orthod. 2022 Jan 25;44(1):86-94. doi: 10.1093/ejo/cjab026. PMID 34041527